CLINICAL TRIAL: NCT01413607
Title: The Use of Self Retaining Sutures in Open and Laparoscopic Partial Nephrectomy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: There was an error made in recruitment therefore patients were not randomized correctly. This was identified in February 2012 and the study was cancelled.
Sponsor: Ricardo Rendon (Other)
Responsible Party: Sponsor-Investigator, Ricardo Rendon, urologist, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Dalhousieurosrs-2011
Record Dates: First submitted 2011-08-02; First posted 2011-08-10 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Kidney Neoplasms
Keywords: nephrectomy; self retaining sutures; laparoscopy
MeSH Terms: conditions — Kidney Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quill knotless tissue-closure device (Experimental): During partial nephrectomy participants in this group will receive the Quill Knotless Tissue-Closure device (Angiotech Pharmaceuticals) to close the central defect in their kidney.
  Interventions: Device: Quill knotless tissue-closure device
- 2-0 absorbable vicryl suture (Active Comparator): Participants in this group will be receiving traditional 2-0 vicryl sutures (Ethicon) during partial nephrectomy.
  Interventions: Device: 2-0 absorbable vicryl suture

INTERVENTIONS:
Device: Quill knotless tissue-closure device — The Quill knotless tissue-closure device is a barbed suture that allows the surgeon to keep tissue approximation without maintaining tension on the suture.
  Other Names: Quill Knotless Tissue-Closure Device (RA-1000Q)
  Arms: Quill knotless tissue-closure device
Device: 2-0 absorbable vicryl suture — In the control group a traditional 2-0 absorbable vicryl suture (Ethicon) will be used to close the central defect in the kidney.
  Other Names: Ethicon 2-0 absorbable vicryl suture
  Arms: 2-0 absorbable vicryl suture

SUMMARY:
The objective of this study is to assess whether using a different type of suture (barbed sutures) during partial nephrectomy results in fewer postoperative complications than with traditional sutures (non-barbed). The most common complications are urine leakage and bleeding. The investigators believe the barbed suture is less technically difficult to use and will allow the surgeon to better repair the hole left in the kidney after the tumor is removed.

DETAILED DESCRIPTION:
With the increased use of radiographic imaging for abdominal complaints the incidental finding of small asymptomatic renal masses has increased. Partial nephrectomy has become the gold standard therapy for treatment of kidney masses ≤7cm in size. Absolute indications for partial nephrectomy include bilateral renal tumors, systemic condition affecting renal function, chronic renal insufficiency and solitary kidney function. Elective indications include masses ≤7cm and normal contralateral kidney function. The procedure can be completed through either laparoscopic or open technique. Complication rates from open and partial nephrectomy have been reported to be about 16% with the most common being urinary leak, postoperative bleeding, renal insufficiency and the need for dialysis.

A major predictor of postoperative complications is the warm ischemia time. This is the length of time the kidney is without blood flow at body temperature. It has been reported that renal and cellular damage of the nephron begins after 20-30 minutes of ischemia. As well, the volume of estimated blood loss has been shown to be a major predictor of postoperative complications. A threshold value of estimated blood loss >750 mL and warm ischemia time >45 minutes have been associated with significantly increased rates of postoperative complications. Recent advancements in laparoscopic technique have lead to the development of the early unclamping method of partial nephrectomy. In this method the renal pedicle is unclamped following the initial central running suture but before the defect has been entirely repaired with bolstering sutures. This method has been reported to decrease warm ischemia time by ≥50% in comparison to the traditional technique of unclamping after full closure of the defect.

The investigators have demonstrated the safety of the "Quill" (Angiotech, Vancouver, BC) polydioxanone barbed self retaining sutures in a retrospective series. These sutures contain unidirectionally oriented barbs on the surface that switch direction at the half-way point. Laparoscopic partial nephrectomy is a technically demanding procedure and maintaining tension during intracorporeal suturing is particularly challenging. The barbs of the self retaining sutures lock into the tissue allowing the surgeon to preserve tissue approximation without needing to maintain tension. The investigators believe these sutures will allow the surgeon to obtain greater tissue approximation therefore decreasing postoperative urinary leakage and bleeding. These findings need to be validated postoperatively.

The investigators believe that coupling the shorter warm ischemia time of the early unclamping method and the greater tissue approximation afforded by the self retaining sutures will result in fewer complications following partial nephrectomy.

ELIGIBILITY:
Inclusion Criteria:

* any person who is being treated for kidney cancer with partial nephrectomy.

Exclusion Criteria:

* those from whom we cannot obtain adequate informed consent.
* those that are converted from partial to radical nephrectomy intraoperatively.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Postoperative bleeding | Data will be collected up to 12 weeks following the procedure
  Patients will be considered positive for bleeding if they have any of gross hematuria, need for transfusion in the postoperative period not believed to be from intraoperative bleeding or need for angioembolization.
Urinary leakage | Data will be collected up to 12 weeks following the procedure
  Urinary leakage is defined as any leakage requiring instrumentation (stent insertion, retrograde pyelogram or percutaneous drainage) or prolonged stay of drain due to high output (>4 days).

SECONDARY OUTCOMES:
Warm or cold ischemia time. | Intraoperative
  Warm is ischemia time is the time that the kidney is without blood perfusion while at body temperature. Cold ischemia time is the time the kidney is without blood perfusion while being cooled below body temperature.
Total operative time | Intraoperative
Length of hospital stay measured in days | Postoperative. Average stay following partial nephrectomy is 3 days
Estimated blood loss during the procedure | Intraoperative

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Rendon, MD, Principal Investigator — Capital distrcit health authority, Canada
Locations (1):
- CDHA QEII site, Halifax, Nova Scotia, Canada

REFERENCES:
- [Background] Becker F, Siemer S, Kamradt J, Zwergel U, Stockle M. Important aspects of organ-preserving surgery for renal tumors: indications, new standards, and oncological outcomes. Dtsch Arztebl Int. 2009 Feb;106(8):117-22. doi: 10.3238/arztebl.2009.0117. Epub 2009 Feb 20. PMID 19568369
- [Background] Becker F, Van Poppel H, Hakenberg OW, Stief C, Gill I, Guazzoni G, Montorsi F, Russo P, Stockle M. Assessing the impact of ischaemia time during partial nephrectomy. Eur Urol. 2009 Oct;56(4):625-34. doi: 10.1016/j.eururo.2009.07.016. Epub 2009 Jul 28. PMID 19656615
- [Background] Gill IS, Kavoussi LR, Lane BR, Blute ML, Babineau D, Colombo JR Jr, Frank I, Permpongkosol S, Weight CJ, Kaouk JH, Kattan MW, Novick AC. Comparison of 1,800 laparoscopic and open partial nephrectomies for single renal tumors. J Urol. 2007 Jul;178(1):41-6. doi: 10.1016/j.juro.2007.03.038. Epub 2007 May 11. PMID 17574056
- [Background] Nguyen MM, Gill IS. Halving ischemia time during laparoscopic partial nephrectomy. J Urol. 2008 Feb;179(2):627-32; discussion 632. doi: 10.1016/j.juro.2007.09.086. Epub 2007 Dec 21. PMID 18082215
- [Background] Turna B, Frota R, Kamoi K, Lin YC, Aron M, Desai MM, Kaouk JH, Gill IS. Risk factor analysis of postoperative complications in laparoscopic partial nephrectomy. J Urol. 2008 Apr;179(4):1289-94; discussion 1294-5. doi: 10.1016/j.juro.2007.11.070. Epub 2008 Mar 4. PMID 18289584
- [Background] El-Ghazaly, T.H. and Rendon, R.A. 2011. Perioperative outcomes of laparoscopic partial nephrectomy using self-retaining sutures (SRS) and early clamp removal versus conventional kidney and collecting system repair. Canadian Urological Association Journal 5(3 suppl 1) s3-s114 sub-article 66